CLINICAL TRIAL: NCT05599984
Title: A Phase 1 First-in-Human Study Evaluating Safety, Pharmacokinetics and Efficacy of ABBV-706 as Monotherapy and in Combination With Budigalimab (ABBV-181), Carboplatin, or Cisplatin in Adult Subjects With Advanced Solid Tumors
Brief Title: Study to Evaluate Adverse Events, Change in Disease Activity, and How ABBV-706 Moves Through the Body When Intravenously (IV) Infused Alone or in Combination With IV Infused Budigalimab, Cisplatin, or Carboplatin in Adult Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M23-385
Record Dates: First submitted 2022-10-28; First posted 2022-10-31 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Small Cell Lung Cancer; Central Nervous System Tumors; ABBV-706; ABBV-181; Budigalimab; Platinum Chemotherapy Combination; Carboplatin; Cisplatin; Neuroendocrine Carcinomas; Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Central Nervous System Neoplasms; Carcinoma, Neuroendocrine; Neoplasms | interventions — Cisplatin; budigalimab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1: ABBV-706 Monotherapy Dose Escalation (Experimental): Participants will receive escalating doses of ABBV-706 until doses for optimization are determined, as part of an approximately 1 year treatment period.
  Interventions: Drug: ABBV-706
- Part 2: ABBV-706 Monotherapy Dose Optimization and Expansion (Experimental): Participants with small cell lung cancer will receive varying doses of ABBV-706 in a randomized manner until the recommended phase 2 dose (RP2D) is achieved, as part of an approximately 1 year treatment period..
  Interventions: Drug: ABBV-706
- Part 3a: ABBV-706 + Budigalimab (Experimental): Participants will receive ABBV-706 in combination with budigalimab, as part of an approximately 1 year treatment period.
  Interventions: Drug: ABBV-706; Drug: Budigalimab
- Part 3b: ABBV-706 + Platinum Chemotherapy (Experimental): Participants will receive ABBV-706 in combination with carboplatin or cisplatin, as part of an approximately 1 year treatment period.
  Interventions: Drug: ABBV-706; Drug: Cisplatin; Drug: Carboplatin
- Part 4a: ABBV-706 Monotherapy Dose Expansion CNS Tumors (Experimental): Participants with relapsed/refractory (R/R) central nervous system (CNS) tumors will receive ABBV-706 as a monotherapy at or below the maximum tolerated dose (MTD) maximum administered dose (MAD), as part of an approximately 1 year treatment period.
  Interventions: Drug: ABBV-706
- Part 4b: ABBV-706 Monotherapy Dose Expansion NECs (Experimental): Participants with R/R neuroendocrine carcinomas (NECs) will receive IV Infused ABBV-706 as a monotherapy at or below the MTD/MAD, as part of an approximately 1 year treatment period.
  Interventions: Drug: ABBV-706

INTERVENTIONS:
Drug: ABBV-706 — Intravenous (IV) Infusion
Drug: Cisplatin — Intravenous infusion
  Arms: Part 3b: ABBV-706 + Platinum Chemotherapy
Drug: Budigalimab — IV Infusion
  Other Names: ABBV-181
  Arms: Part 3a: ABBV-706 + Budigalimab
Drug: Carboplatin — Intravenous infusion
  Arms: Part 3b: ABBV-706 + Platinum Chemotherapy

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess safety, tolerability, pharmacokinetics and preliminary efficacy of ABBV-706 as a monotherapy and in combination with budigalimab, carboplatin, or cisplatin.

ABBV-706 is an investigational drug being developed for the treatment of small cell lung cancer (SCLC), high-grade central nervous system (CNS) tumors and high-grade neuroendocrine carcinomas (NECs). There are multiple treatment arms in this study. Participants will either receive ABBV-706 as a single agent or in combination with budigalimab (another investigational drug), carboplatin or cisplatin at different doses. Approximately 350 adult participants will be enrolled in the study across sites worldwide.

In part 1 (dose escalation), ABBV-706 will be intravenously infused in escalating doses as a monotherapy until the maximum tolerated dose (MTD) is determined in participants with SCLC, high-grade CNS tumors, and high-grade NECs. In part 2, multiple doses will be selected from Part 1 and SCLC participants will be assigned to one of these doses in a randomized fashion to determine the recommended Phase 2 dose. In Part 3a, participants with SCLC or NECs will receive ABBV-706 in combination with budigalimab intravenously every 3 weeks. In Part 3b participants with SCLC or NECs will receive ABBV-706 in combination with either carboplatin or cisplatin intravenously. In Part 4a, participants with CNS tumors will receive ABBV-706 intravenously at a dose determined from Part 1. In Part 4b, participants with NECs will receive ABBV-706 intravenously at a dose selected from Part 1. The estimated duration of the study is up to 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The laboratory values criteria must be met within 7 days prior to the first dose of study drug as per the protocol.
* QT interval corrected for heart rate (QTc) <= 450 msec (males) or <= 470 msec (females) using Fridericia's correction, and an ejection fraction of >= 50% as measured by echocardiogram or multigated acquisition (MUGA) scan at Screening.
* Part 1 only: Advanced recurrent or refractory solid tumors with potential SEZ6 expression including small cell lung cancer (SCLC), high-grade central nervous system (CNS) tumors (glioblastoma [GBM], IDH-wildtype Grade 4; oligodendroglioma, IDH-mutant, and 1p/19q-codeleted Grade 3; astrocytoma, IDH-mutant Grade 3 or Grade 4), neuroendocrine prostate cancer (NEPC), high-grade poorly differentiated gastroenteropancreatic neuroendocrine carcinoma (GEP-NEC)s, large cell neuroendocrine carcinoma (LCNEC)s, SCLC transformed from epidermal growth factor receptor (EGFR) mutant non-small cell lung cancer (NSCLC), atypical lung carcinoids, and other high-grade poorly differentiated NECs, who have progressed on or after standard of care (SoC) therapy and with no curative therapy available. For SCLC, participants must have histologically or cytologically confirmed SCLC that is relapsed or refractory following at least 1 prior platinum-containing chemotherapy.
* Part 2 only: Histologically or cytologically confirmed SCLC that is relapsed or refractory (R/R) following at least 1 prior platinum-containing chemotherapy and with no curative therapy available. For the purposes of this study, a line of therapy is defined as >= 1 complete cycle of either a single agent or combination of drugs, including any planned sequential therapy of various regimens.
* Part 3a only: Participants with R/R SCLC following at least 1 prior platinum-containing chemotherapy or R/R poorly differentiated NECs, e.g., NEPC, GEP-NECs, LCNECs, SCLC transformed from EGFR mutant Non-small cell lung cancer (NSCLC), atypical lung carcinoids, other high-grade poorly differentiated NECs.
* Part 3b only: Participants with R/R SCLC who have only progressed following a frontline regimen containing a platinum-based chemotherapy or R/R NECs, e.g., NEPC, GEP-NECs, LCNECs, SCLC transformed from EGFR mutant NSCLC, atypical lung carcinoids, other NECs.
* Part 4a only: Participants with R/R high-grade CNS tumors (GBM, IDH-wildtype Grade 4; oligodendroglioma, IDH-mutant, and 1p/19q-codeleted Grade 3; astrocytoma, IDH-mutant Grade 3 or Grade 4) who have progressed on SoC therapy and with no curative therapy options available.
* Part 4b only: Participants with R/R neuroendocrine tumors, including NEPC, GEP-NECs, LCNECs, SCLC transformed from EGFR mutant NSCLC, atypical lung carcinoids, and other high-grade poorly differentiated NECs, who have progressed on SoC therapy and with no curative therapy options available.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for participants with extracranial solid tumors or Response Assessment for Neuro-Oncology (RANO)for participants with primary high-grade CNS tumors (GBM, IDH-wildtype Grade 4; oligodendroglioma, IDH-mutant, and 1p/19q-codeleted Grade 3; astrocytoma, IDH-mutant Grade 3 or Grade 4).
* Primary CNS tumors within 12 weeks from radiation therapy should have unequivocal progression as documented by either tumor recurrence predominantly outside of radiation field on magnetic resonance imaging (MRI) or confirmed on tumor biopsy.
* Participants with brain metastases from an extracranial solid tumor are eligible if the brain metastases as outlined in the protocol.
* Fresh or archival tumor tissue available for submission, for retrospective SEZ6 expression analysis as outlined in the protocol.

Exclusion Criteria:

* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, nor any evidence of active ILD or pneumonitis.
* History of idiopathic pulmonary fibrosis or organizing pneumonia.
* Prior treatment with an antibody drug conjugate that consists of a Top1 inhibitor payload.
* Part 2 only: Prior treatment with a SEZ6-targeted antibody drug conjugate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AE) | Up to Approximately 2 Years
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum/Plasma Concentration (Cmax) of ABBV-706 | Up to Approximately 2 Years
  Maximum observed serum/plasma concentration of ABBV-706.
Time to Cmax (Tmax) of ABBV-706 | Up to Approximately 2 Years
  Time to Cmax of ABBV-706.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-706 | Up to Approximately 2 Years
  Terminal phase elimination half-life (t1/2) of ABBV-706.
Area Under the Serum/Plasma Concentration-Time Curve (AUC) of ABBV-706 | Up to Approximately 2 Years
  Area under the serum/plasma concentration-time curve of ABBV-706.
Antidrug Antibodies (ADAs) | Up to Approximately 2 Years
  Incidence and concentration of anti-drug antibodies.
Neutralizing Antibodies (nAbs) | Up to Approximately 2 Years
  Incidence and concentration of neutralizing antibodies.
Percentage of Participants with Objective Response, for Participants with Extracranial Solid Tumors | Up to Approximately 2 Years
  Objective response is defined as participants achieving a confirmed best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 for for extracranial solid tumors per investigator assessment.
Recommended Phase 2 Dose (RP2D) of ABBV-706 | Up to Approximately 2 Years
  The RP2D will be determined using all available information, including, but not limited to, AEs, dose-limiting toxicities, pharmacokinetic parameters, clinical laboratory tests, and efficacy measures.
Percentage of Participants with Objective Response for Participants with Central Nervous System (CNS) Tumors | Up to Approximately 2 Years
  Objective response is as participants achieving a confirmed best overall response of CR and PR according to Response Assessment for Neuro-Oncology (RANO), version 1.1 for CNS tumors per investigator assessment.
Duration of response (DOR) for Participants with Confirmed CR/PR | Up to Approximately 2 Years
  For participants achieving a confirmed CR/PR, DOR is defined as the time from the initial response of CR/PR to disease progression or death of any cause, whichever occurs earlier.
Percentage of Participants with Clinical Benefit | Up to Approximately 2 Years
  Clinical benefit is defined as a participant achieving CR/PR, or Stable Disease (SD).
Progression-Free Survival (PFS) | Up to Approximately 2 Years
  PFS is defined as time from first study treatment to a documented disease progression, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Overall survival (OS) | Up to Approximately 2 Years
  OS is defined as time from first study treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (66):
- United States (22):
  - Banner MD Anderson Cancer Ctr /ID# 260129, Gilbert, Arizona
  - City Of Hope Comprehensive Cancer Center /ID# 271295, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 259884, Irvine, California
  - Yale New Haven Hospital /ID# 246647, New Haven, Connecticut
  - Georgetown University Hospital /ID# 255352, Washington D.C., District of Columbia
  - University of Chicago Medical Center /ID# 256334, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc /ID# 260130, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics /ID# 246638, Iowa City, Iowa
  - Barbara Ann Karmanos Cancer In /ID# 261799, Detroit, Michigan
  - Henry Ford Hospital /ID# 246648, Detroit, Michigan
  - START Midwest /ID# 251257, Grand Rapids, Michigan
  - St. Lukes Hosp. of Kansas City /ID# 259958, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 246286, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 246303, New York, New York
  - Duke Cancer Center /ID# 246285, Durham, North Carolina
  - UH Cleveland Medical Center /ID# 246641, Cleveland, Ohio
  - Univ Oklahoma HSC /ID# 250884, Oklahoma City, Oklahoma
  - Tennessee Oncology, PLLC /ID# 246283, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center /ID# 246287, Houston, Texas
  - South Texas Accelerated Research Therapeutics /ID# 248946, San Antonio, Texas
  - University of Utah /ID# 246640, Salt Lake City, Utah
  - Northwest Medical Specialties - Tacoma /ID# 262801, Tacoma, Washington
- Australia (4):
  - Chris O'Brien Lifehouse /ID# 259087, Camperdown, New South Wales
  - The Kinghorn Cancer Centre /ID# 260874, Darlinghurst, New South Wales
  - Austin Health and Ludwig Institute for Cancer Research /ID# 255174, Heidelberg, Victoria
  - Peter MacCallum Cancer Ctr /ID# 259197, Melbourne, Victoria
- China (6):
  - Cancer Hospital - Chinese Academy Of Medical Sciences /ID# 270044, Beijing, Beijing Municipality
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 270038, Wuhan, Hubei
  - First Affiliated Hospital of China Medical University /ID# 270041, Shenyang, Liaoning
  - Shanghai Chest Hospital /ID# 270036, Shanghai, Shanghai Municipality
  - Shanghai East Hospital /ID# 268615, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital /Id# 270039, Shanghai, Shanghai Municipality
- France (3):
  - Institut Bergonie /ID# 258655, Bordeaux, Gironde
  - Institut Gustave Roussy /ID# 260334, Villejuif, Val-de-Marne
  - Institut Régional du Cancer Montpellier /ID# 265086, Montpellier
- Germany (3):
  - Klinikum der Universitaet Muenchen - Campus Innenstadt /ID# 259412, Munich, Bavaria
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 259414, Dresden, Saxony
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin /ID# 259413, Berlin
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 254915, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 255059, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 255147, Jerusalem
- Italy (2):
  - Istituto Europeo Di Oncologia /ID# 256804, Milan, Milano
  - Fondazione IRCCS San Gerardo dei Tintori - Ospedale San Gerardo /ID# 258228, Monza, Monza E Brianza
- Japan (8):
  - National Cancer Center Hospital East /ID# 259417, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center /ID# 261279, Matsuyama, Ehime
  - Hokkaido Cancer Center /ID# 261278, Sapporo, Hokkaido
  - Kyoto University Hospital /ID# 259419, Kyoto, Kyoto
  - Shizuoka Cancer Center /ID# 261277, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 259418, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 260132, Koto-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 260131, Wakayama, Wakayama
- South Korea (6):
  - National Cancer Center /ID# 248938, Goyang-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 248939, Seongnam, Gyeonggido
  - Chonnam National University Hwasun Hospital /ID# 248943, Hwasun-gun, Jeonranamdo
  - Seoul National University Hospital /ID# 248940, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 248936, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 248937, Seoul
- Spain (9):
  - Hospital HM Nou Delfos /ID# 264851, Barcelona
  - Hospital Universitario Vall de Hebron /ID# 258659, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 257294, Barcelona
  - Hospital Universitario Ramon y Cajal /ID# 257291, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 257295, Madrid
  - Hospital Universitario 12 de Octubre /ID# 258658, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 258657, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 256940, Seville
  - Hospital Clinico Universitario de Valencia /ID# 257290, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-108